CLINICAL TRIAL: NCT04167501
Title: Impact of HPV Vaccination on the Distribution of HPV in High Grade Lesions of the Cervix in France
Brief Title: Impact of HPV Vaccination on Cervical High Grade Lesions in France
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/454
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2020-07

CONDITIONS: Human Papillomavirus Infection
Keywords: cervical precancerous lesion; HPV; vaccination; Impact study; France
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non exposed: Women born between 1972 and 1982 who were not exposed to HPV vaccination
  Interventions: Other: biological sample analysis
- exposed: Women born between 1983 and 1993 who were potentially exposed to HPV vaccination
  Interventions: Other: biological sample analysis

INTERVENTIONS:
Other: biological sample analysis — HPV Prevalence analysis

SUMMARY:
The objective is to estimate the prevalence of the different genotypes of human papillomaviruses (HPV) in histologically proven high-grade lesions of the cervix in patients born between 1972 and 1993. It is plan to determine if the prevalence of HPV16 and HPV18 is lower in the population born between 1983 and 1993 and potentially exposed to HPV vaccination compared to those born between 1972 and 1982 who were not exposed to vaccination. Thus the investigators should be able to determine whether the introduction of HPV vaccination in France in 2007 has had an impact on the development of high-grade lesions associated with HPV16 and HPV18.

DETAILED DESCRIPTION:
The prevalence of the different HPV in high-grade lesions (CIN2/3) will be determined using the INNOLiPA HPV extra v2 genotyping kit (Fujirebio). Only samples with a histologically proven high-grade cervical lesion (grade 2 or 3 intraepithelial neoplasia) are concerned. The patient year of birth, the year of the lesion diagnosis and the histological diagnosis will be recorded Participating laboratories will select eligible cervical samples (biopsies or surgical specimen) according to the inclusion criteria defined in the protocol. Only cervical samples with sufficient biological material will be selected. The selected tissue blocks will be sent to the Papillomavirus National Reference Center (NRC) by mail (pre-paid envelope provided) in accordance with the rules for the transport of biological samples. After receipt by the NRC, the tissue blocks will be anonymized. After HPV genotyping, the blocks will be returned to the laboratory. Transport costs are covered by the Papillomavirus NRC.

Samples have to be fixed in 4% buffered formaldehyde (maximum 24 hours) and then included in paraffin for histopathological evaluation. On each of the selected histological pieces, the papillomavirus NRC will make 5μm thick sections using a microtome. The number of sections to be made depends on the size of the histological specimen. A minimum surface area equivalent to 5 sections of 5μm of a 125 mm2 piece is required for genotyping.

Tissue sections are grouped in a labelled 2 mL screw tube. To avoid any contamination between samples, the microtome blade will be carefully cleaned with xylene and then 95% ethanol between each block.

After DNA extraction using the QiaAmp DNA mini Kit (Qiagen), HPV genotype analysis will be performed using molecular techniques for the detection of human papillomavirus DNA. The investigators will use the INNO-LiPA HPV Genotyping Extra II (Fujirebio) kit. This is a Polymerase Chain Reaction (PCR) technique using degenerate primers followed by reverse hybridization on strips on which the specific probes of 32 alpha HPV genotypes are immobilized. This kit allows the detection of 13 high-risk HPV genotypes (HPV16, 18, 31, 33, 35, 39, 45, 51, 52, 52, 56, 58, 59, 68), 6 HPVs that are likely to be at risk (HPV 26, 53, 66, 70, 73, 82) and 14 low-risk or unclassified HPVs (HPV6, 11, 40, 42, 43, 44, 54, 61, 62, 67, 81, 83, 89). In addition, the samples will be analyzed by PCR luminex according to the technique published by Schmitt et al, J Clin Microbiol 2010. In addition to alpha HPV, this technique allows the detection of sixty beta and gamma HPVs.

Characteristics of the subjects to be included A description of patients included in the study (women born between 1972 and 1982, on the one hand, and women born between 1983 and 1993, on the other) will include age at time of sampling, year of sampling, stage of lesion CIN2 or 3, and histological type.

Comparisons between age groups will be made using Student tests for quantitative variables and Chi-square tests for qualitative variables, while respecting the conditions for applying these tests.

Main judgment criteria Prevalences of high-risk HPV 16 or 18 genotypes will be described in both age groups with their 95% confidence intervals. These prevalences will be compared between the two age groups using the Chi-square test.

Secondary Judgment Criterion Prevalences of high-risk HPV genotypes other than 16 or 18 will be described in both age groups with their 95% confidence intervals. These prevalences will be compared between the two age groups using the Chi-square test.

Additional analyses The distribution of the different HPV genotypes will be described for both age groups.

The number of samples required for the study is 606: 303 samples from women born between 1972 and 1982 and 303 samples from women born between 1983 and 1993.

The calculation of the number of samples required is based on the following assumptions: the prevalence of HPV16 and/or HPV18 in high-grade lesions of women is estimated at 62%. The minimum decrease after the introduction of HPV vaccination, interesting from a population health point of view, that the investigators wish to highlight is 10%, i.e. an expected prevalence among women born between 1983 and 1993 of 52%.

For a power set at 80% and an alpha risk at 5%, a unilateral formulation of hypotheses (only a decrease in prevalence is possible) and an equal number of samples from women aged 25-34 and 35-44, the number of samples required per group is 303.

ELIGIBILITY:
Inclusion Criteria:

* High grade lesions of the cervix
* Histologic diagnosis of cervical intraepithelial neoplasia grade 2 or 3, carinoma in situ
* Biopsy or surgical specimen
* Formalin-fixed ans paraffin embedded specimen

Exclusion Criteria:

- samples fixed in Boin's solution

Ages: 27 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women born between 1972 and 1993
Sampling Method: Probability Sample
Enrollment: 606 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
HPV16 and HPV18 prevalence | 18 months
  Prevalence of HPV16 and HPV18 genotypes in high grade cervical lesions of the cervix in women born between 1972 and 1993

SECONDARY OUTCOMES:
Other HPV prevalence | 18 months
  Prevalence of high risk HPV other than HPV16 and HPV18 genotypes and prevalence of low risk HPV in high grade cervical lesions of the cervix in women born between 1972 and 1993

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc PRETET, Pr, Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (1):
- CHU Besançon, Besançon, France

REFERENCES:
- [Derived] Lenoir P, Guillet J, Desmarets M, Baraquin A, Ramanah R, Rousse J, Mougin C, Lepiller Q, Pretet JL; HPV Impact Study Group. Human papillomavirus genotype distribution among high-grade cervical lesions in French women born between 1972 and 1993. J Gynecol Obstet Hum Reprod. 2025 May;54(5):102945. doi: 10.1016/j.jogoh.2025.102945. Epub 2025 Mar 21. PMID 40122237